CLINICAL TRIAL: NCT03169894
Title: Phase Ib Escalating Dose, Open-Label, Signal-Finding Study to Evaluate the Safety, Tolerability, and Short-Term Efficacy of the Anti-Light Monoclonal Antibody MDGN-002 in Adults With Moderate to Severe Active Crohn's Disease or Ulcerative Colitis Who Previously Failed Treatment With an Anti-TNFα Agent
Brief Title: Evaluation of the Safety, Tolerability, and Efficacy of MDGN-002 in Adults With Moderate to Severe Active Crohn's Disease or Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic reasons
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDGN-002-CD-101
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-07

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MDGN-002 (Experimental): MDGN-002 will be supplied in vials of 150 mg/mL. MDGN-002 will be administered by SQ injection in the abdomen every 14 days at 1 of 2 dose levels: 1.0 mg/kg or 3.0 mg/kg.
  Interventions: Drug: MDGN-002

INTERVENTIONS:
Drug: MDGN-002 — MDGN-002 is a fully human IgG4 monoclonal antibody specific to human LIGHT.
  Other Names: AVTX-002, AEVI-002

SUMMARY:
This is a Phase 1b, open-label, dose-escalation, signal-finding, multi-center study. The study will evaluate the safety, tolerability, pharmacokinetics and short-term efficacy of MDGN-002 in adults with moderate to severe, active Crohn's disease or Ulcerative Colitis who have previously failed anti-tumor necrosis factor alpha (anti-TNFα) treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, ≥ 18 to ≤ 75 years of age.
2. Subject has a documented diagnosis of CD via endoscopy/colonoscopy and histological confirmation, or subject has received a diagnosis of UC for 90 days or greater prior to Visit 1, confirmed by endoscopy during the Screening Period, with exclusion of current infection, dysplasia and/or malignancy.
3. Subject has moderate to severe, active CD as evidenced Simple Endoscopy Score for Crohn's Disease (SES-CD) score of ≥7, and histological confirmation, or subject has moderately to severely active UC, as defined by a Modified Mayo Score (excluding the PGA component) of 5 to 9 points at Visit 1.
4. Subject has failed treatment with an approved therapeutic dose of an anti-TNFα monoclonal antibody treatment.

Exclusion Criteria:

1. Subject has a diagnosis of ulcerative colitis (UC) or indeterminate colitis or subject has a diagnosis of Crohn's disease or indeterminate colitis .
2. Subject with signs or symptoms of bowel obstruction.
3. Subject has short bowel syndrome.
4. Subject has a current functional colostomy or ileostomy.
5. Subject has had a surgical bowel resection within the past 6 months prior to screening or is planning any resection during the study period.
6. Subject is pregnant or a nursing mother.
7. Subject is sexually active and not using effective contraception as defined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Sweet Hope Research Specialty, Inc., Hialeah, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Egleston Hospital, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Hassman Research Institute, Berlin, New Jersey
  - University of Cincinnati, Cincinnati, Ohio
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - The Center for Pediatric Inflammatory Bowel Disease, Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC, San Antonio, Texas
  - Care Access Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: MDGN-002 1.0 mg/kg
- Cohort 2: MDGN-002 3.0 mg/kg
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 4 | 4
Safety Analysis Set | 4 | 4
Full Analysis Set | 4 | 4
PK Analysis Set | 4 | 3
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (14.66) | 26.5 (5.07) | 35.9 (14.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Population: BMI not available for all subjects
  kg/m2
    number analyzed (Participants) | 4 | 3 | 7
    (all) | 27.37 (10.192) | 15.84 (4.428) | 22.43 (9.820)
Time Since Diagnosis (Years) [Mean (Standard Deviation); unit: years] | 25.2 (6.17) | 6.2 (2.18) | 15.7 (11.00)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD)
Description: The SES-CD is assessed through endoscopic review of 5 predefined gastrointestinal (GI) segments (ileum; right colon; transverse colon; left colon; rectum). For each segment, 4 endoscopic variables are assessed (presence of ulcers, ulcerated surface, affected surface, and presence of narrowing). Each variable is scored from 0 to 3 with higher scores indicating more severe symptoms. For each variable, the total score is calculated as the sum across all segments of the GI tract. The SES-CD total score, ranging from 0-60, is calculated as the sum of all variable total scores with a higher score indicating more severe endoscopic activity
Time Frame: Baseline to Visit 10 (Day 56) or early termination
Population: Full Analysis Set, with data analyzed and presented only for subjects with both a Baseline and Visit 10 or Early Termination assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 4
score on a scale | -4.0 (4.36) | 1.3 (7.50)

2. Secondary Outcome: Change From Baseline in Crohn's Disease Activity Index (CDAI)
Description: The Crohn's Disease Activity Index (CDAI) consists of the following 8 items: abdominal pain, number of liquid stools, general well-being, extraintestinal complication, use of antidiarrheal drugs, abdominal mass, hematocrit, and body weight. Information on abdominal pain, general well-being, and frequency of loose and watery stools was taken from a daily diary completed by the subject.
  Total CDAI scores can range from 0 to approximately 600 with higher scores indicating more active disease. Disease severity as measured by CDAI is categorized as: Remission (<150), Mildly active disease (150 - 219); Moderately active disease (220 - 450); Severe disease (> 450).
Time Frame: Baseline to Visit 10 (Day 56) or early termination.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 1
score on a scale | -19.2 (38.34) | -123.6 (NA) — a standard deviation cannot be calculated for a single measure.

3. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBD-Q).
Description: The IBD-Q is a 32-item questionnaire validated to measure quality of life in Crohn's disease subjects. The IBD-Q assesses the dimensions of bowel function, emotional status, systemic symptoms, and social function.
  Each of the 32 items is scored on a 1 to 7 scale, where higher scores represent a more positive response, and better outcome. The IBD-Q total score is calculated as the sum of all 32 items in the questionnaire, ranging from 32 to 224.
Time Frame: Baseline to Visit 10 (Day 56) or Early Termination
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
score on a scale | 43.5 (29.01) | 47.0 (31.59)

4. Secondary Outcome: Change From Baseline in Total Number of Stools Daily
Description: Subjects reported their daily stool frequency including loose and/or watery stools via a diary. The stool frequency including the number of loose and/or watery stools per day, equivalent to a score of a 6 or 7 on the Bristol Stool Scale, was recorded. Loose stools were described as fluffy pieces with ragged edges, a mushy stool. Watery stools were described as watery, no solid pieces.
Time Frame: Baseline to Visit 10 (Day 56) or Early Termination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of total daily stools
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 2
number of total daily stools | 1.37 (0.286) | -0.99 (4.462)

5. Secondary Outcome: Change From Baseline in Total Number of Loose/Watery Stools Daily
Description: Subjects reported their daily assessment of stool frequency including loose and/or watery stools via a diary. The stool frequency including the number of loose and/or watery stools per day, equivalent to a score of a 6 or 7 on the Bristol Stool Scale, was recorded. Loose stools were described as fluffy pieces with ragged edges, a mushy stool. Watery stools were described as watery, no solid pieces.
Time Frame: Baseline to Visit 10 (Day 56) or Early Termination
Population: Full Analysis Set with data analyzed and presented only for subjects with both a Baseline and Visit 10 or Early Termination assessment
Measure: Mean (Standard Deviation); unit: number of daily loose/watery stools
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 2
number of daily loose/watery stools | 0.90 (1.077) | -1.07 (5.758)

6. Secondary Outcome: Change From Baseline in Abdominal Pain
Description: Subjects reported their daily assessment of abdominal pain via a diary. Abdominal pain was assessed on a scale of 0 to 3 with higher values indicating greater pain severity.
Time Frame: Baseline to Visit 10 (Day 56) or Early Termination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 2
score on a scale | -0.75 (0.354) | 0.18 (0.455)

7. Secondary Outcome: Change From Baseline in General Well-Being
Description: Subjects reported their daily assessment of well-being via a diary. General well being was assessed on a scale of 0 to 4, with higher values indicating a poorer condition of health.
Time Frame: Baseline to Visit 10 (Day 56) or Early Termination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 2 | 2
score on a scale | -0.11 (0.859) | -0.27 (0.623)

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the time of the informed consent until the final safety follow-up visit (Day 84 or 28 days after Early Termination). This included events occurring during the screening phase of the study, regardless of whether investigational product was administered. Therefore all serious and non-serious events are included regardless of meeting or not meeting the study definition of treatment emergent.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/4
Other Adverse Events (participants affected / at risk) | 2/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=4)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Tunnel vision (Nervous system disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an open label study, exploratory in nature, without a placebo control group, and as such, limits the interpretation of the study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03169894/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT03169894/SAP_001.pdf